CLINICAL TRIAL: NCT00006159
Title: Family-Centered Diabetes Project for Pueblo Native Americans
Brief Title: Family-Centered Diabetes Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Purpose: Treatment
Other Study IDs: carterj (completed); R01DK047096 (NIH)
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes
Keywords: diabetes; lifestyle intervention; Native American; community intervention; diet; exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise; Diet; Community Support

INTERVENTIONS:
Behavioral: lifestyle (exercise, diet, and family and community support)

SUMMARY:
The purpose of this project is to determine whether a diabetes lifestyle program will improve the lives of Native American people living with diabetes. We recruited Native American people living in 8 Pueblo communities served by 3 Indian Health Service clinics. Forty percent of people living with diabetes in those communities participated in an interview and had height, weight, blood pressure and hemoglobin A1c measured at the beginning. Then they received a lifestyle program in either groups or one-on-one, or another group which got the intervention after one year (comparison group). The program was developed using input from community members, tribal leaders, and clinic staff, and was taught by community members in or near the participating communities. After each session, participants were asked for feedback about the curriculum. After the program ended, the interview and clinical measures were repeated. Feedback to tribal leaders and clinical staff is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older with diabetes living in a participating Native American community served by one of three participating Indian Health Service clinics.

Exclusion Criteria:

* Unable to complete a yearly interviewer administered questionnaire and clinical measures of height, weight, blood pressure, and fingerstick hemoglobin A1c.
* Unable to participate in 5 lifestyle intervention meetings occurring over a one year period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-03; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janette S. Carter, MD, Principal Investigator — University of New Mexico School of Medicine
Locations (1):
- University of New Mexico School of Medicine, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Gilliland SS, Carter JS, Perez GE, Two Feathers J, Kenui CK, Mau MK. Recommendations for development and adaptation of culturally competent community health interventions in minority populations with Type 2 diabetes mellitus. Diabetes Spectrum 11:166-174, 1998.
- [Background] McFee T, Cunningham-Sabo LD, Perez GE, Gilliland SS, Carter JS. A feast day poster: Healthful and successful modification of holiday foods. J Nutr Educ 29:356B, 1997. (two page ''GEM'' article)
- [Background] Stolarczyk LM, Gilliland SS, Lium DJ, Owen CL, Perez GE, Kriska AM, Ainsworth BE, Carter JS. Knowledge, attitudes and behaviors related to physical activity among Native Americans with diabetes. Ethn Dis. 1999 Winter;9(1):59-69. PMID 10355475
- [Background] Carter JS, Pugh JA, Monterrosa A. Non-insulin-dependent diabetes mellitus in minorities in the United States. Ann Intern Med. 1996 Aug 1;125(3):221-32. doi: 10.7326/0003-4819-125-3-199608010-00011. PMID 8686981
- [Background] Carter JS, Wiggins CL, Becker TM, Key CR, Samet JM. Diabetes mortality among New Mexico's American Indian, Hispanic, and non-Hispanic white populations, 1958-1987. Diabetes Care. 1993 Jan;16(1):306-9. doi: 10.2337/diacare.16.1.306. PMID 8422797
- [Background] Carter J, Horowitz R, Wilson R, Sava S, Sinnock P, Gohdes D. Tribal differences in diabetes: prevalence among American Indians in New Mexico. Public Health Rep. 1989 Nov-Dec;104(6):665-9. PMID 2511603
- [Background] Carter JS, Gilliland SS, Perez GE, Skipper B, Gilliland FD. Public health and clinical implications of high hemoglobin A1c levels and weight in younger adult Native American people with diabetes. Arch Intern Med. 2000 Dec 11-25;160(22):3471-6. doi: 10.1001/archinte.160.22.3471. PMID 11112241
- [Background] Griffin JA, Gilliland SS, Perez G, Helitzer D, Carter JS. Participant satisfaction with a culturally appropriate diabetes education program: the Native American Diabetes Project. Diabetes Educ. 1999 May-Jun;25(3):351-63. doi: 10.1177/014572179902500306. PMID 10531855
- [Background] Griffin JA, Gilliland SS, Perez G, Upson D, Carter JS. Challenges to participating in a lifestyle intervention program: the Native American Diabetes Project. Diabetes Educ. 2000 Jul-Aug;26(4):681-9. doi: 10.1177/014572170002600416. PMID 11140076
- [Background] Carter JS, Perez GE, Gilliland SS. Communicating through stories: experience of the Native American Diabetes Project. Diabetes Educ. 1999 Mar-Apr;25(2):179-88. doi: 10.1177/014572179902500204. PMID 10531844
- [Background] Gilliland SS, Willmer AJ, McCalman R, Davis SM, Hickey ME, Perez GE, Owen CL, Carter JS. Adaptation of the Dartmouth COOP Charts for use among American Indian people with diabetes. Diabetes Care. 1998 May;21(5):770-6. doi: 10.2337/diacare.21.5.770. PMID 9589238
- [Background] Carter JS, Houston CA, Gilliland SS, Perez GE, Owen CL, Pathak DR, Little RR. Rapid HbA1c testing in a community setting. Diabetes Care. 1996 Jul;19(7):764-7. doi: 10.2337/diacare.19.7.764. PMID 8799636
- [Background] Gilliland FD, Owen C, Gilliland SS, Carter JS. Temporal trends in diabetes mortality among American Indians and Hispanics in New Mexico: birth cohort and period effects. Am J Epidemiol. 1997 Mar 1;145(5):422-31. doi: 10.1093/oxfordjournals.aje.a009124. PMID 9048516
- [Background] Carter JS, Gilliland SS, Perez GE, Levin S, Broussard BA, Valdez L, Cunningham-Sabo LD, Davis SM. Native American Diabetes Project: designing culturally relevant education materials. Diabetes Educ. 1997 Mar-Apr;23(2):133-4, 139. doi: 10.1177/014572179702300203. No abstract available. PMID 9155311
- See also: The intervention curricula, Strong in Body and Spirit! (participant version) is located at this web site and may be downloaded. — http://www.laplaza.org/health/dwc/prof/nadp/